CLINICAL TRIAL: NCT04601350
Title: Effect of Remimazolam Use During Perioperative Period on Brain Waves and Postoperative Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20200922
Record Dates: First submitted 2020-10-05; First posted 2020-10-23 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Benzodiazepine
Keywords: remimazolam; recovery
MeSH Terms: interventions — remimazolam; Anesthesia, General; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam 1 (Experimental)
  Interventions: Drug: remimazolam group was induced with remimazolam 0.1 mg/kg followed by a maintenance dose of 0.1 mg·kg-1·h-1 for general anesthesia
- Control (Other)
  Interventions: Drug: control group was induced with midazolam 0.05 mg/kg followed by normal saline maintenance of 0.1 ml·kg-1·h-1

INTERVENTIONS:
Drug: remimazolam group was induced with remimazolam 0.1 mg/kg followed by a maintenance dose of 0.1 mg·kg-1·h-1 for general anesthesia — remimazolam group was remimazolam 0.1 mg/kg followed by a maintenance dose of 0.1 mg·kg-1·h-1 for general anesthesia
  Arms: Remimazolam 1
Drug: control group was induced with midazolam 0.05 mg/kg followed by normal saline maintenance of 0.1 ml·kg-1·h-1 — control group was induced with midazolam 0.05 mg/kg followed by normal saline maintenance of 0.1 ml·kg-1·h-1
  Arms: Control

SUMMARY:
Benzodiazepine sedative hypnotics are commonly used intravenous anesthetics in clinical practice. Remimazolam is a new benzodiazepine with the characteristics of rapid onset, short maintenance and recovery time, no accumulation, metabolism independent of liver and kidney function, and no serious side effects, which has a good prospect for clinical application. Now we will study the effects of remimazolam on EEG and postoperative cognitive function ，in order to further understand the clinical application of remimazolam.

ELIGIBILITY:
Inclusion Criteria:

* ASAⅠ-Ⅱ
* Patients undergoing elective surgery under general anesthesia.
* Age, sex, and weight were not limited.

Exclusion Criteria:

* Allergic or contraindication to remimazolam/midazolam/remifentanil;
* Abnormal liver and kidney function; Alcohol abuse;
* Long-term use of sedative, analgesic or anxiolytic drugs;
* Hearing and language communication disorders;
* Complicated with severe cardiovascular lesions or neurological diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The average intraoperative power spectral density in the frontal alpha band | Preoperatively, During operation，End of operation
  EEG data were collected at the beginning of the room admission, and the collection was ended at the end of the operation.
Changes in the score of MMSE | The outcome above should be measured the day before surgery and 1,2,3,5,7 days after surgery
  The outcome above should be measured the day before surgery and 1,2,3,5,7 days after surgery

SECONDARY OUTCOMES:
Changes in IL-6, IL-10, and S100-β levels | The outcome above should be measured the day before surgery and 1，3 days after surgery
  The outcome above should be measured the day before surgery and 1，3 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China